CLINICAL TRIAL: NCT06031493
Title: A Multimodal Intervention Program to Improve Sexual Health and Self-perceived Quality of Life in Patients Treated for Cervical Cancer: a Randomized Prospective Study (PROVIDENCE Trial)
Brief Title: A Multimodal Intervention Program to Improve Sexual Health and Self-perceived Quality of Life in Patients Treated for Cervical Cancer (PROVIDENCE)
Acronym: PROVIDENCE
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hospital Clinic of Barcelona (Other)
Collaborators: Hospital Universitario 12 de Octubre (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PROVIDENCE
Record Dates: First submitted 2023-09-04; First posted 2023-09-11 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2023-08

CONDITIONS: Cervical Cancer; Sexual Dysfunction; Quality of Life
Keywords: cervical cancer; sexual dysfunction
MeSH Terms: conditions — Uterine Cervical Neoplasms; Sexual Dysfunction, Physiological | interventions — Quality of Life

STUDY DESIGN:
Intervention Model Description: prospective, multi-institutional, national, randomized clinical trial with two parallel arms.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Multimodal Intervention Group (Experimental): Multimodal Intervention on sexual dysfunction and quality-of-life after treatment for cervical cancer: application of topical vaginal estrogens, systematic evaluation of the need of systemic hormone replacement therapy (and treatment if needed), application of hormone-free vaginal-vulvar moisturizing cream containing hyaluronic acid, use of a vaginal vibrator twice a week for 5 to 10 minutes each time with the help of intimate lubricant, access to online informational content about sexuality, access to online informational content about nutrition, access to online informational content about sports, access to online informational content about lifestyle habits
  Interventions: Combination Product: Multimodal intervention on sexual dysfunction and quality-of-life
- Standard Care Group (No Intervention): Standard follow-up in Gynecological Oncology Units of participating centers after treatment for cervical cancer

INTERVENTIONS:
Combination Product: Multimodal intervention on sexual dysfunction and quality-of-life — Multimodal intervention includes education on healthy habits, the prevention of vaginal dysfunction using vaginal moisturizers and topical estrogens, and a systematic evaluation of the need of hormone replacement therapy.
  Arms: Multimodal Intervention Group

SUMMARY:
The PROVIDENCE Trial aims to explore the improvement of sexual health and self-perceived health related quality of life (measured by Patient Reported Outcome Measures) through a multimodal intervention that includes patient education on healthy habits and the prevention of vaginal dysfunction using vaginal moisturizers and topical estrogens. To achieve this, a randomized design is proposed to assess sexual health and quality of life in patients treated for cervical cancer who undergo this intervention compared to those who receive standard care.

DETAILED DESCRIPTION:
Cervical cancer treatment, both radical hysterectomy and chemoradiotherapy, can impair all scopes of daily life and, beyond the physical changes caused by treatment, has psychological and social implications that influence health-related quality of life (HR-QoL). Patients undergoing treatment for cervical cancer have shown to score less in HR-QoL scales compared to healthy women. More than half of women with gynecological cancer experience sexual dysfunction, especially those affected by cervical cancer. In spite of the latest 2023 ESGO/ESTRO/ESP recommendations on the management of cervical cancer, several observational studies indicate that the percentage of cervical cancer patients receiving information and treatment for early menopause and sexual dysfunction, especially regarding hormone replacement therapy, does not exceed 50%.

The PROVIDENCE trial is a multi-institutional, national, randomized clinical trial which aims to demonstrate that a multimodal intervention including patient education on sexuality and healthy habits and the prevention of vaginal dysfunction reduces sexual disfunction and HR-QoL impairment in patients treated for cervical cancer. The recruitment period is scheduled from January 2024 to December 2026 and will be held in Gynecology Oncology Units of referral hospitals in Spain.

Patients will be randomized 1:1 at diagnosis of cervical cancer to control arm or intervention arm. After treatment for initial or locally advanced cervical cancer, patients in the control arm will undergo the standard follow-up and treatment of post-treatment morbidity will be performed following the standard procedures as determined by their referring physician. The proposed multimodal intervention for patients assigned to the intervention group (detailed below) includes education on healthy habits, the prevention of vaginal dysfunction using vaginal moisturizers and topical estrogens, and a systematic evaluation of the need of hormone replacement therapy.

ELIGIBILITY:
Inclusion Criteria:

* Women older that 18 years, with initial or locally advanced primary cervical cancer
* Squamous, adenocarcinoma or adenosquamous histology
* Stage I-III cervical cancer treated with surgery and/or radiotherapy ± systemic treatment in - Gynecology Oncology Units of referral hospitals in Spain
* Signed informed consent by the patient or legal guardian

Exclusion Criteria:

* Women younger tan 18 years
* Pregnancy or breastfeeding
* Patients with intraepithelial lesions of cervix uteri without invasive disease
* Metastatic tumor in the cervix uteri or primary tumor with atypical histology
* Inability to complete the questionnaires included in the study protocol
* Contraindications for the use of topical vaginal estrogens
* Patients undergoing fertility-preservation treatment (conization or trachelectomy)
* Patients undergoing palliative treatment

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 122 (Estimated)
Dates: Start 2025-01 (Estimated); Primary Completion 2025-02 (Estimated); Study Completion 2025-04 (Estimated)

PRIMARY OUTCOMES:
FSFI score | 12 months after completion of primary treatment for cervical cancer
  global score in FSFI (Female Sexual Function Index) questionnaire

SECONDARY OUTCOMES:
FSFI (6 months) | 6 months after completion of primary treatment for cervical cancer
  global score in FSFI (Female Sexual Function Index) questionnaire
EORTC QLQ-30 | 12 months after completion of primary treatment for cervical cancer
  global score in EORTC (European Organisation for Research and Treatment of Cancer) QLQ-30 questionnaire
EORTC QLQ-30 (6 months) | 6 months after completion of primary treatment for cervical cancer
  global score in EORTC QLQ-30 questionnaire
EORTC Cx-24 (6 months) | 6 months after completion of primary treatment for cervical cancer
  global score in EORTC Cx-24 questionnaire
EORTC Cx-24 | 12 months after completion of primary treatment for cervical cancer
  global score in EORTC Cx-24 questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Blanca Gil-Ibáñez, MD, PhD, Study Director — Hospital Universitario 12 de Octubre; Berta Díaz-Feijoo, MD, PhD, Study Director — Hospital Clinic of Barcelona
Locations (2):
- Spain (2):
  - Hospital Clínic de Barcelona, Barcelona
  - Hospital Universitario 12 de Octubre, Madrid

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Gil-Ibanez B, Carreras-Dieguez N, Lopez G, Sanchez-Hoyo B, Nuno BC, Oliver-Perez R, Castelo-Branco C, Marina T, Torne A, Tejerizo A, Diaz-Feijoo B. A multimodal intervention program to improve sexual health and self-perceived quality of life in patients treated for cervical cancer: a randomized prospective study (PROVIDENCE trial). J Gynecol Oncol. 2025 Jul;36(4):e56. doi: 10.3802/jgo.2025.36.e56. Epub 2025 Jan 29. PMID 39924671